CLINICAL TRIAL: NCT02612909
Title: A Phase 2/3 Double Blinded, Randomized, Placebo-controlled Study in Healthy Adult Volunteers in Vietnam to Examine the Safety and Immunogenicity of an Inactivated A/H5N1 Influenza Vaccine (IVACFLU-A/H5N1) Produced by IVAC
Brief Title: A Safety and Immunogenicity Study of IVACFLU-A/H5N1
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Institute of Vaccines and Medical Biologicals, Vietnam (Industry)
Collaborators: National Institute of Hygiene and Epidemiology, Vietnam (Other); World Health Organization (Other); Department of Health and Human Services (U.S. Federal Agency); PATH (Other); FHI 360 (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: IVACFLU-A/H5N1-0203; NCT02815098 (obsolete NCT alias)
Record Dates: First submitted 2015-10-15; First posted 2015-11-24 (Estimated); Results first posted 2019-04-16 (Actual); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: Avian Influenza
Keywords: Avian Influenza; A/H5N1 vaccine; IVAC
MeSH Terms: conditions — Influenza in Birds

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Phase 2: Placebo (Placebo Comparator): Subjects participating in Phase 2 and assigned to receiving two injections of placebo administered intramuscularly as a single dose, separated by 21 days.
  Interventions: Biological: Placebo
- Phase 2: Vaccine (15 mcg) (Active Comparator): Subjects participating in Phase 2 and assigned to receiving two injections of IVACFLU-A/H5N1 vaccine (15 mcg concentration) administered intramuscularly as a single dose, separated by 21 days.
  Interventions: Biological: IVACFLU-A/H5N1 vaccine
- Phase 2: Vaccine (30 mcg) (Active Comparator): Subjects participating in Phase 2 and assigned to receiving two injections of IVACFLU-A/H5N1 vaccine (30 mcg concentration) administered intramuscularly as a single dose, separated by 21 days.
  Interventions: Biological: IVACFLU-A/H5N1 vaccine
- Phase 3: Placebo (Placebo Comparator): Subjects participating in Phase 3 and assigned to receiving two injections of placebo administered intramuscularly as a single dose, separated by 21 days.
  Interventions: Biological: Placebo
- Phase 3: Vaccine (Experimental): Subjects participating in Phase 2 and assigned to receiving two injections of IVACFLU-A/H5N1 vaccine (15 mcg concentration) administered intramuscularly as a single dose, separated by 21 days.
  Interventions: Biological: IVACFLU-A/H5N1 vaccine

INTERVENTIONS:
Biological: IVACFLU-A/H5N1 vaccine — Monovalent A/H5N1 influenza vaccine (MIV), whole virion inactivated, purified by sucrose gradient on ultracentrifuge. The vaccine was produced in eggs, inactivated with formaldehyde, and formulated with aluminum hydroxide 0.6 mg/0.5 mL with no preservative.
  Arms: Phase 2: Vaccine (15 mcg); Phase 2: Vaccine (30 mcg); Phase 3: Vaccine
Biological: Placebo — Includes 4.500mg sodium chloride, 0.685 mg sodium phosphate dibasic dihydrate, and 0.186 mg sodium phosphate monobasic dihydrate.
  Other Names: Sterile Phosphate Buffered Saline (PBS)
  Arms: Phase 2: Placebo; Phase 3: Placebo

SUMMARY:
The study hypothesis was that two 0.5 mL doses of whole virion monovalent A/H5N1 influenza vaccine (IVACFLU-A/H5N1) adjuvanted with alum would be safe and well tolerated in healthy adults, and that at least one of the two doses tested would be immunogenic in 60% or more of the subjects tested.

DETAILED DESCRIPTION:
Although the A/H1N1 (2009) pandemic has subsided and the virus has become endemic, the threat of another pandemic due to avian influenza A/H5N1 remains constant. Since 1997, highly pathogenic A/H5N1 avian viruses have caused both widespread outbreaks in poultry with high mortality and sporadic, severe, and fatal disease in humans. Southeast Asian countries, including Vietnam, have been affected by influenza A/H5N1. From 2003 through March 2015, WHO has reported 826 confirmed human cases of A/H5N1 influenza infection; including 440 fatal cases (World Health Organization, 2015). Southeast Asian countries accounted for 42% of all confirmed influenza A/H5N1 cases reported since 2003, and influenza A/H5N1 infection in animals is now thought to be endemic in the region (World Health Organization, 2015). As of March 2015, Vietnam has reported 127 confirmed human cases and 64 deaths. In 2014, two cases of A/H5N1 avian influenza were reported in Vietnam. Therefore, the risk of transmission to human is still present.

At the time of the study, no influenza A/H5N1 vaccine had been licensed in Vietnam. IVACFLU-A/H5N1 is an influenza A/H5N1 vaccine produced by Institute of Vaccines and Medical Biologicals (IVAC) using embryonated chicken eggs. IVACFLU-A/H5N1 is a whole virus vaccine, collected in a linear sucrose density gradient solution using a continuous flow centrifuge (Alfa Wassermann, West Caldwell, NJ) and inactivated with formaldehyde. The vaccine is alum adjuvanted. Vaccine strain NIBRG-14 derived from original influenza A/Vietnam/1194/2004 was provided to IVAC by the National Institute for Biological Standards and Control of the Health Protection Agency of the United Kingdom. A clinical trial of IVACFLU-A/H5N1 vaccine conducted in 75 subjects at the Ben Luc Health District in Vietnam in 2014 showed that the vaccine is safe and immunogenic at doses of 7.5 and 15 mcg.

This study was conducted in two stages: Phase 2 was a dose selection study where subjects were randomized to one of the three groups (15 mcg IVACFLU-A/H5N1 vaccine, 30 mcg IVACFLU-A/H5N1 vaccine or placebo) at a 1:1:1 ratio. The conduct of Phase 3 was dependent on showing hemagglutination inhibition (HAI) response titer of ≥1:40 in ≥60% of vaccine recipients in at least one of the two Phase 2 IVACFLU-A/H5N1 vaccine groups. Based on the review of immunogenicity and safety results from the Phase 2 study, a dose of study vaccine was selected for Phase 3. Subjects were randomized at two sites (Khanh Hoa and Hai Phong) to receive the IVACFLU-A/H5N1 vaccine dose selected in Phase 2 or placebo . Safety was assessed in all subjects and immunogenicity was measured in a subset of subjects at the Hai Phong study site.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adult 18 through 60 years of age at the enrollment visit.
* Literate (by self-report) and willing to provide written informed consent.
* Healthy adults, as established by the medical history and screening evaluations, including physical examination, capable and willing to complete Diary Cards, and willing to return for all follow-up visits.
* For females able to become pregnant, willing to utilize reliable birth control measures (intrauterine device, hormonal contraception, condoms) through the Day 43 visit.

Exclusion Criteria:

* Participation in another clinical trial involving any vaccine or therapy within the previous three months, or planned enrollment in such a trial during the period of this study.
* Received any non-study vaccine within 4 weeks prior to enrollment or refused to postpone receipt of such vaccines until after the Day 43 visit.
* Current or recent (within 2 weeks of enrollment) acute illness with or without fever.
* Received immune globulin or other blood products within 3 months prior to study enrollment or planned receipt of such products prior to the Day 43 visit.
* Chronic administration (defined as more than 14 consecutively-prescribed days) of immunosuppressants or other immune-modulating therapy within six months prior to study enrollment. (For corticosteroids, this meant prednisone or equivalent, 0.5 mg per kg per day; topical or intranasal steroids were allowed.)
* History of asthma.
* Hypersensitivity after previous administration of any vaccine.
* Suspected or known hypersensitivity to any of the study vaccine components, including chicken or egg protein, antibiotics, and rubber (from the vaccine vial stoppers).
* Acute or chronic clinically significant pulmonary, cardiovascular, hepatobiliary, metabolic, neurologic, psychiatric, or renal functional abnormality, as determined by medical history, physical examination, or clinical laboratory screening tests (Phase 2 only), which in the opinion of the investigator, might have interfered with the study objectives.
* History of any blood or solid organ cancer.
* History of thrombocytopenic purpura or known bleeding disorder.
* History of seizures.
* Known or suspected immunosuppressed or immune deficient condition of any kind.
* Known Hepatitis B Virus (HBV) or Hepatitis C virus (HCV) infection by self-report (Phase 3) or a positive test for either HBV surface antigen (HBsAg) or HCV antibody using anti-HCV test (Phase 2).
* Known HIV infection (self-report)
* Known active tuberculosis or symptoms of active tuberculosis (self-report).
* History of chronic alcohol abuse and/or illegal drug use.
* Pregnancy or lactation (a negative pregnancy test was required before administration of study product for all women of childbearing potential).
* History of Guillain-Barre Syndrome.
* Any condition in the opinion of the investigator that would have increased the health risk of the subject if he/she participated in the study or interfered with the evaluation of the study objectives.

Note: Minor out-of-range laboratory values no greater than Grade 1 were not considered to be exclusionary at screening.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 930 (Actual)
Dates: Start 2017-03-07 (Actual); Primary Completion 2017-08-29 (Actual); Study Completion 2017-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tran N Duong, MD, PhD, Principal Investigator — National Institute of Hygiene and Epidemiology, Vietnam
Locations (2):
- Vietnam (2):
  - Phase 3: Hai Phong Provincial Preventive Medicine Center, Haiphong, Hai Phong
  - Phase 2 & 3: Khanh Hoa Provincial Health Department, Nha Trang, Khanh Hoa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Duong TN, Thiem VD, Anh DD, Cuong NP, Thang TC, Huong VM, Chien VC, Phuong NTL, Montomoli E, Holt R, Scorza FB, Flores J, Tewari T. A Phase 2/3 double blinded, randomized, placebo-controlled study in healthy adult participants in Vietnam to examine the safety and immunogenicity of an inactivated whole virion, alum adjuvanted, A(H5N1) influenza vaccine (IVACFLU-A/H5N1). Vaccine. 2020 Feb 5;38(6):1541-1550. doi: 10.1016/j.vaccine.2019.11.059. Epub 2019 Dec 4. PMID 31812464

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Phase 2 & 3: Recruitment occurred from communes affiliated with the District Health Centers. Commune health workers identified potential participants through home visits and invited interested people to attend an information session. People heard about the study and those interested had individual consent for screening.
Groups:
- Phase 3: Vaccine: Subjects participating in Phase 3 and assigned to receiving two injections of IVACFLU-A/H5N1 vaccine (15 mcg concentration) administered intramuscularly as a single dose, separated by 21 days.
Period: Phase 2
Arm/Group | Phase 2: Placebo | Phase 2: Vaccine (15 mcg) | Phase 2: Vaccine (30 mcg) | Phase 3: Placebo | Phase 3: Vaccine
Started | 100 | 100 | 100 | 0 | 0
Received Injection 1 | 100 | 100 | 100 | 0 | 0
Received Injection 2 | 98 | 95 | 99 | 0 | 0
Completed Day 29 Clinic Visit (8 days after injection 2) | 98 | 95 | 99 | 0 | 0
Completed Day 43 Clinic Visit (22 days after injection 2 (immunogenicity assessed)) | 97 | 94 | 99 | 0 | 0
Completed | 98 | 95 | 99 | 0 | 0
Not Completed | 2 | 5 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 5 | 0 | 0 | 0
Not completed — Pregnancy | 0 | 0 | 1 | 0 | 0
Period: Phase 3
Arm/Group | Phase 2: Placebo | Phase 2: Vaccine (15 mcg) | Phase 2: Vaccine (30 mcg) | Phase 3: Placebo | Phase 3: Vaccine
Started | 0 | 0 | 0 | 105 | 525
Received Injection 1 | 0 | 0 | 0 | 105 | 525
Received Injection 2 | 0 | 0 | 0 | 103 | 520
Completed Day 29 Clinic Visit | 0 | 0 | 0 | 104 | 525
Completed Day 43 Clinic Visit | 0 | 0 | 0 | 104 | 524
Completed | 0 | 0 | 0 | 104 | 525
Not Completed | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 2: Placebo | Phase 2: Vaccine (15 mcg) | Phase 2: Vaccine (30 mcg) | Phase 3: Placebo | Phase 3: Vaccine | Total
Number analyzed (Participants) | 100 | 100 | 100 | 105 | 525 | 930
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.6 (9.62) | 39.8 (9.99) | 39.7 (9.63) | 39.9 (9.61) | 40.2 (9.72) | 40.0 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 72 | 65 | 66 | 286 | 550
  Male | 39 | 28 | 35 | 39 | 239 | 380
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Kinh | 100 | 100 | 100 | 105 | 524 | 929
  Other | 0 | 0 | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number and Percentage of Subjects Achieving a Hemagglutination Inhibition (HAI) Titer of ≥1:40
Description: Serum specimens were tested for the presence of HAI antibodies to influenza. The HAI assay was conducted using serum samples from all the subjects in Phase 2 of the study and in a subset of approximately 270 subjects receiving the IVACFLU-A/H5N1 vaccine (vaccinees) and placebo from one study site in Phase 3 in order to have at least 200 evaluable subjects receiving IVACFLU-A/H5N1 and 40 evaluable subjects receiving placebo, at the end of study.
Time Frame: Day 1, Day 43
Population: Subjects who received 2 injections and had valid sera samples for the day measured
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: Placebo | Phase 2: Vaccine (15 mcg) | Phase 2: Vaccine (30 mcg) | Phase 3: Placebo | Phase 3: Vaccine
Number analyzed (Participants) | 98 | 95 | 99 | 45 | 222
Participants
  Day 1 | 0 | 0 | 0 | 0 | 1
  Day 43: number analyzed (Participants) | 97 | 95 | 99 | 45 | 222
  Day 43 | 0 | 79 | 81 | 0 | 98

2. Secondary Outcome: Phase 2: Number and Percentage of Subjects Achieving a Hemagglutination Inhibition (HAI) Titer of ≥1:40
Description: as for outcome 1
Time Frame: Day 1, Day 22
Population: Subjects who received 2 injections and had valid sera samples for the day measured
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: Placebo | Phase 2: Vaccine (15 mcg) | Phase 2: Vaccine (30 mcg)
Number analyzed (Participants) | 98 | 95 | 99
Participants
  Day 1 | 0 | 0 | 0
  Day 22 | 0 | 42 | 56

3. Secondary Outcome: Phase 2: Number and Percentage of Subjects Achieving at Least a 4-fold Increase in Hemagglutination Inhibition (HAI) Titer
Description: Serum specimens were tested for the presence of HAI antibodies to influenza on day 1, day 22, and day 43 (day 1 and 22 prior to injection). The HAI assay was conducted using serum samples from all the subjects in Phase 2 of the study and in a subset of approximately 270 subjects receiving the IVACFLU-A/H5N1 vaccine (vaccinees) and placebo from one study site in Phase 3 in order to have at least 200 evaluable subjects receiving IVACFLU-A/H5N1 and 40 evaluable subjects receiving placebo, at the end of study.
Time Frame: Day 22, Day 43
Population: Subjects who received the prior injections (as applicable) and had valid sera samples for the day measured
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: Placebo | Phase 2: Vaccine (15 mcg) | Phase 2: Vaccine (30 mcg)
Number analyzed (Participants) | 98 | 95 | 99
Participants
  Day 22 | 0 | 57 | 70
  Day 43 | 0 | 88 | 93

4. Secondary Outcome: Phase 3: Number and Percentage of Subjects Achieving at Least a 4-fold Increase in Hemagglutination Inhibition (HAI) Titer
Description: as for outcome 1
Time Frame: Day 43
Population: Subjects who received 2 injections and had valid sera samples for the day measured
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 3: Placebo | Phase 3: Vaccine
Number analyzed (Participants) | 45 | 222
Participants | 0 | 150

5. Secondary Outcome: Phase 2: Geometric Mean Hemagglutination Inhibition (HAI) Titer
Description: as for outcome 3
Time Frame: Day 1, Day 22, Day 43
Population: Subjects who received the prior injections (as applicable) and had valid sera samples for the day measured
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Phase 2: Placebo | Phase 2: Vaccine (15 mcg) | Phase 2: Vaccine (30 mcg)
Number analyzed (Participants) | 98 | 95 | 99
titer
  Day 1 | 5.48 [5.23 to 5.74] | 5.62 [5.34 to 5.91] | 5.68 [5.30 to 6.10]
  Day 22 | 5.52 [5.26 to 5.80] | 31.67 [24.60 to 40.77] | 42.16 [33.45 to 53.13]
  Day 43: number analyzed (Participants) | 97 | 95 | 99
  Day 43 | 5.63 [5.31 to 5.96] | 62.65 [52.10 to 75.34] | 59.20 [49.87 to 70.28]

6. Secondary Outcome: Phase 3: Geometric Mean Hemagglutination Inhibition (HAI) Titer
Description: as for outcome 1
Time Frame: Day 1, Day 43
Population: Subjects who received 2 injections and had valid sera samples for the day measured
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Phase 3: Placebo | Phase 3: Vaccine
Number analyzed (Participants) | 45 | 222
titer
  Day 1 | 5.04 [4.96 to 5.11] | 5.08 [4.97 to 5.18]
  Day 43 | 5.20 [5.06 to 5.34] | 27.61 [24.38 to 31.27]

7. Secondary Outcome: Phase 2: Geometric Mean Hemagglutination Inhibition (HAI) Titer Ratio, With Respect to Day 1
Description: as for outcome 3
Time Frame: Day 22, Day 43
Population: Subjects who received the prior injections (as applicable) and had valid sera samples for the day measured
Measure: Geometric Mean (95% Confidence Interval); unit: fold change
Arm/Group | Phase 2: Placebo | Phase 2: Vaccine (15 mcg) | Phase 2: Vaccine (30 mcg)
Number analyzed (Participants) | 98 | 95 | 99
fold change
  Day 22 | 1.01 [0.99 to 1.02] | 5.64 [4.43 to 7.18] | 7.42 [5.93 to 9.27]
  Day 43: number analyzed (Participants) | 97 | 95 | 99
  Day 43 | 1.03 [1.00 to 1.05] | 11.15 [9.35 to 13.29] | 10.41 [8.79 to 12.34]

8. Secondary Outcome: Phase 3: Geometric Mean Hemagglutination Inhibition (HAI) Titer Ratio, With Respect to Day 1
Description: as for outcome 1
Time Frame: Day 43
Population: Subjects who received 2 injections and had valid sera samples for the day measured
Measure: Geometric Mean (95% Confidence Interval); unit: fold change
Arm/Group | Phase 3: Placebo | Phase 3: Vaccine
Number analyzed (Participants) | 45 | 222
fold change | 1.01 [0.99 to 1.02] | 5.31 [4.69 to 6.02]

9. Secondary Outcome: Number and Percentage of Subjects Experiencing Reactogenicity
Description: Immediate reactogenicity (30 minutes post-injection) were evaluated on Day 1 and Day 22 and consisted of:
  * Inspection of the upper arms for the presence or absence of redness, swelling, hardness, pain, or tenderness; and
  * Documentation of the presence or absence of headache, fever, fatigue/malaise, muscle aches, joint aches, nausea, vomiting, or chills.
  Immediate reactogenicity were assessed by a study physician or appropriately trained medical staff.
Time Frame: 30 minutes after each injection
Population: Subjects who received injections
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: Placebo | Phase 2: Vaccine (15 mcg) | Phase 2: Vaccine (30 mcg) | Phase 3: Placebo | Phase 3: Vaccine
Number analyzed (Participants) | 100 | 100 | 100 | 105 | 525
Participants
  Injection 1: any local reaction | 0 | 1 | 1 | 0 | 1
  Injection 1: any systemic reaction | 1 | 1 | 0 | 0 | 0
  Injection 2: any local reaction: number analyzed (Participants) | 98 | 95 | 99 | 105 | 525
  Injection 2: any local reaction | 2 | 2 | 2 | 2 | 3
  Injection 2: any systemic reaction: number analyzed (Participants) | 98 | 95 | 99 | 105 | 525
  Injection 2: any systemic reaction | 0 | 1 | 0 | 2 | 2

10. Secondary Outcome: Number and Percentage of Subjects Experiencing Reactogenicity
Description: Reported solicited signs and symptoms were recorded by the subject on the Diary Card from Days 1-7 and Days 22-28 in the study, then evaluated by study physician on Days 8, 22, and 29.The evaluated solicited local reactogenicity events were as follows:
  * Size of redness (at site of injection) in centimeters (cm)
  * Size of swelling (at site of injection) in cm
  * Size of induration (hardness at site of injection) in cm
  * Pain (at site of injection)
  * Tenderness (at site of injection)
  The evaluated solicited systemic reactogenicity events were as follows:
  * Fever/body temperature (and body location of measurement)
  * Fatigue/malaise
  * Generalized muscle aches
  * Joint aches/pains
  * Chills
  * Nausea
  * Vomiting
  * Headache
Time Frame: 7 days after each vaccination
Population: Subjects who received injections
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: Placebo | Phase 2: Vaccine (15 mcg) | Phase 2: Vaccine (30 mcg) | Phase 3: Placebo | Phase 3: Vaccine
Number analyzed (Participants) | 100 | 100 | 100 | 105 | 525
Participants
  Injection 1: any local reaction | 22 | 83 | 87 | 19 | 409
  Injection 1: any systemic reaction | 52 | 66 | 83 | 36 | 286
  Injection 2: any local reaction: number analyzed (Participants) | 98 | 95 | 99 | 103 | 520
  Injection 2: any local reaction | 12 | 44 | 50 | 15 | 227
  Injection 2: any systemic reaction: number analyzed (Participants) | 98 | 95 | 99 | 103 | 520
  Injection 2: any systemic reaction | 29 | 31 | 37 | 19 | 129

11. Secondary Outcome: Number and Percentage of Subjects Experiencing Unsolicited Adverse Events (AE)
Description: Unsolicited AEs were any AEs that occurred any time after study product was given (temporally related to study product), whether or not deemed "related" to the product, and were not solicited. Unsolicited AEs were either observed by study staff while the subject was at a clinic for a study visit or reported by the subject at any time. Any solicited sign or symptom starting after 7 days post-study product injection was recorded as an "unsolicited AE".
  For the Phase 2 study, laboratory results were considered AEs when the result was Grade 2 or above.
  Any medical condition that was present at the time that the subject was enrolled was not reported as an AE, but was reported as a pre-existing condition on the Medical History Form. However, if this condition occurred with greater frequency or severity during the study, it was recorded as an AE.
Time Frame: 21 days after each vaccination
Population: Subjects who received injections
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: Placebo | Phase 2: Vaccine (15 mcg) | Phase 2: Vaccine (30 mcg) | Phase 3: Placebo | Phase 3: Vaccine
Number analyzed (Participants) | 100 | 100 | 100 | 105 | 525
Participants
  Injection 1: at least one AE | 21 | 20 | 24 | 16 | 73
  Injection 1: at least 1 severe AE | 3 | 0 | 0 | 0 | 0
  Injection 1: at least 1 treatment-related AE | 1 | 0 | 1 | 0 | 0
  Injection 2: at least one AE: number analyzed (Participants) | 98 | 95 | 99 | 103 | 520
  Injection 2: at least one AE | 6 | 10 | 11 | 16 | 56
  Injection 2: at least 1 severe AE: number analyzed (Participants) | 98 | 95 | 99 | 103 | 520
  Injection 2: at least 1 severe AE | 1 | 2 | 1 | 1 | 0
  Injection 2: at least 1 treatment-related AE: number analyzed (Participants) | 98 | 95 | 99 | 103 | 520
  Injection 2: at least 1 treatment-related AE | 0 | 0 | 0 | 0 | 0

12. Secondary Outcome: Number and Percentage of Subjects Experiencing Unsolicited Serious Adverse Events (SAE)
Description: Defined as an adverse event that led to death, was life-threatening (subject at immediate risk of death); required inpatient hospitalization or prolongation of existing hospitalization; resulted in congenital anomaly/birth defect; resulted in a persistent or significant disability or incapacity.
Time Frame: 90 days
Population: Subjects who received injections
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: Placebo | Phase 2: Vaccine (15 mcg) | Phase 2: Vaccine (30 mcg) | Phase 3: Placebo | Phase 3: Vaccine
Number analyzed (Participants) | 100 | 100 | 100 | 105 | 525
Participants | 0 | 1 | 0 | 4 | 8

13. Secondary Outcome: Phase 2: Number and Percentage of Subjects Achieving at Least a 4-fold Increase in Neutralizing Antibody Titer
Description: The microneutralization (MN) assay is an alternative assay for determining immunologic response to vaccination. It is a highly sensitive assay that can provide information on the ability of induced antibody to neutralize influenza virus. Titers of neutralizing antibodies were expressed as the amount of the greatest dilution of serum giving a neutralization of 50% of tissue cytopathic effects of the virus in the tissue culture.
Time Frame: Day 22, Day 43
Population: Subjects who received the prior injections (as applicable) and had valid sera samples for the day measured
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: Placebo | Phase 2: Vaccine (15 mcg) | Phase 2: Vaccine (30 mcg)
Number analyzed (Participants) | 98 | 95 | 99
Participants
  Day 22 | 0 | 21 | 26
  Day 43 | 0 | 57 | 63

14. Secondary Outcome: Phase 3: Number and Percentage of Subjects Achieving at Least a 4-fold Increase in Neutralizing Antibody Titer
Description: The MN assay is an alternative assay for determining immunologic response to vaccination. It is a highly sensitive assay that can provide information on the ability of induced antibody to neutralize influenza virus. Titers of neutralizing antibodies were expressed as the amount of the greatest dilution of serum giving a neutralization of 50% of tissue cytopathic effects of the virus in the tissue culture.
  In Phase 3, MN assay was conducted in a subset of approximately 270 subjects receiving the IVACFLU-A/H5N1 vaccine (vaccinees) and placebo from one study site in order to have at least 200 evaluable subjects receiving IVACFLU A/H5N1 and 40 evaluable subjects receiving placebo.
Time Frame: Day 43
Population: Subjects who received 2 injections and had valid sera samples for the day measured
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 3: Placebo | Phase 3: Vaccine
Number analyzed (Participants) | 45 | 222
Participants | 0 | 114

15. Secondary Outcome: Phase 2: Geometric Mean Neutralizing Antibody Titer
Description: as for outcome 13
Time Frame: Day 1, Day 22, Day 43
Population: Subjects who received the prior injections (as applicable) and had valid sera samples for the day measured
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Phase 2: Placebo | Phase 2: Vaccine (15 mcg) | Phase 2: Vaccine (30 mcg)
Number analyzed (Participants) | 98 | 95 | 99
titer
  Day 1 | 7.15 [7.03 to 7.26] | 7.10 [7.04 to 7.15] | 7.19 [7.07 to 7.33]
  Day 22 | 7.12 [7.02 to 7.22] | 13.78 [11.23 to 16.92] | 29.76 [24.47 to 36.20]
  Day 43: number analyzed (Participants) | 97 | 95 | 99
  Day 43 | 7.12 [7.02 to 7.22] | 29.76 [24.47 to 36.20] | 28.48 [24.34 to 33.32]

16. Secondary Outcome: Phase 3: Geometric Mean Neutralizing Antibody Titer
Description: as for outcome 1
Time Frame: Day 1, Day 43
Population: Subjects who received 2 injections and had valid sera samples for the day measured
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Phase 3: Placebo | Phase 3: Vaccine
Number analyzed (Participants) | 45 | 222
titer
  Day 1 | 7.07 [7.07 to 7.07] | 7.07 [7.07 to 7.07]
  Day 43 | 7.07 [7.07 to 7.07] | 26.16 [22.66 to 30.20]

17. Secondary Outcome: Phase 2: Geometric Mean Neutralizing Antibody Titer Ratio, With Respect to Day 1
Description: as for outcome 13
Time Frame: Day 22, Day 43
Population: Subjects who received the prior injections (as applicable) and had valid sera samples for the day measured
Measure: Geometric Mean (95% Confidence Interval); unit: fold change
Arm/Group | Phase 2: Placebo | Phase 2: Vaccine (15 mcg) | Phase 2: Vaccine (30 mcg)
Number analyzed (Participants) | 98 | 95 | 99
fold change
  Day 22 | 1.00 [0.99 to 1.00] | 1.94 [1.59 to 2.38] | 2.02 [1.67 to 2.45]
  Day 43: number analyzed (Participants) | 97 | 95 | 99
  Day 43 | 1.00 [0.99 to 1.00] | 4.19 [3.46 to 5.09] | 3.96 [3.38 to 4.63]

18. Secondary Outcome: Phase 3: Geometric Mean Neutralizing Antibody Titer Ratio, With Respect to Day 1
Description: as for outcome 14
Time Frame: Day 43
Population: Subjects who received 2 injections and had valid sera samples for the day measured
Measure: Geometric Mean (95% Confidence Interval); unit: fold change
Arm/Group | Phase 3: Placebo | Phase 3: Vaccine
Number analyzed (Participants) | 45 | 222
fold change | 1.00 [1.00 to 1.00] | 3.70 [3.21 to 4.27]

ADVERSE EVENTS:
Time Frame: 21 days for non-serious adverse events, 90 days for serious adverse events
Arm/Group | Phase 2: Placebo | Phase 2: Vaccine (15 mcg) | Phase 2: Vaccine (30 mcg) | Phase 3: Placebo | Phase 3: Vaccine
All-Cause Mortality (participants affected / at risk) | 0/100 | 0/100 | 0/100 | 0/105 | 0/525
Serious Adverse Events (participants affected / at risk) | 0/100 | 1/100 | 0/100 | 4/105 | 8/525
Other Adverse Events (participants affected / at risk) | 21/100 | 20/100 | 24/100 | 17/105 | 58/525
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 2: Placebo (N=100) | Phase 2: Vaccine (15 mcg) (N=100) | Phase 2: Vaccine (30 mcg) (N=100) | Phase 3: Placebo (N=105) | Phase 3: Vaccine (N=525)
Abdominal adhesion (Gastrointestinal disorders) | NA | 0 | NA | 0 | 1
Abdominal symptom (Gastrointestinal disorders) | NA | 0 | NA | 1 | 0
Appendicitis (Gastrointestinal disorders) | NA | 0 | NA | 1 | 1
Concussion (Injury, poisoning and procedural complications) | NA | 0 | NA | 0 | 1
Diverticulitis (Gastrointestinal disorders) | NA | 0 | NA | 0 | 1
Electric shock (Injury, poisoning and procedural complications) | NA | 0 | NA | 1 | 1
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | NA | 0 | NA | 1 | 1
Tonsillitis (Respiratory, thoracic and mediastinal disorders) | NA | 1 | NA | 0 | 0
Viral fever (Infections and infestations) | NA | 0 | NA | 0 | 1
Wound (Injury, poisoning and procedural complications) | NA | 0 | NA | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 2: Placebo (N=100) | Phase 2: Vaccine (15 mcg) (N=100) | Phase 2: Vaccine (30 mcg) (N=100) | Phase 3: Placebo (N=105) | Phase 3: Vaccine (N=525)
Insomnia (Nervous system disorders) | 1 | 0 | 1 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 2 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 2 | 1 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Periodontal inflammation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 2 | 2 | 0 | 1
Nasopharyngitis (Infections and infestations) | 3 | 3 | 2 | 0 | 0
Varicella (Infections and infestations) | 0 | 0 | 2 | 0 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0 | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 4 | 1 | 0 | 0 | 0
Blood pressure increased (Investigations) | 1 | 0 | 2 | 0 | 0
White blood cell count increased (Investigations) | 1 | 0 | 2 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 1 | 0 | 0
Headache (Nervous system disorders) | 2 | 1 | 1 | 0 | 0
Vestibular disorder (Nervous system disorders) | 0 | 1 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 1 | 3
Influenza (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 | 5 | 6 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 3 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 4
Skin infection (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 0 | 1
Rhinitis allergic (Immune system disorders) | 1 | 0 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1
Sciatica (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Tonsillitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0
Tooth extraction (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0
Vestibular disorder (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 6
Abdominal symptom (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 2
Aphthous ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Oropharyngeal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Periodontitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Burning sensation (General disorders) | 0 | 0 | 0 | 1 | 0
Inflammation (General disorders) | 0 | 0 | 0 | 0 | 4
Pain (General disorders) | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 2
Urticaria (Immune system disorders) | 0 | 0 | 0 | 1 | 2
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Ear infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 5 | 11
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 3 | 12
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Gastritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Gingivitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Gout (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Headache (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 3
Back pain (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Vertigo (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 3
Calculus urinary (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Laryngitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Herpes Zoster (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 1
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 10
Injection site bruising (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Tricuspid valve incompetence (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 1
Refraction disorder (Eye disorders) | 0 | 0 | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Pharyngitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Cervicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Sebaceous gland infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 2
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Abdominal adhesion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Electric shock (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 6
Neck pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2
Pyelonephritis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Subcutaneous abscess (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2015-12-22): https://cdn.clinicaltrials.gov/large-docs/09/NCT02612909/SAP_000.pdf
  • Study Protocol (2015-11-24): https://cdn.clinicaltrials.gov/large-docs/09/NCT02612909/Prot_001.pdf